CLINICAL TRIAL: NCT01198184
Title: Safety and Efficacy of RO4929097 in Combination With Temsirolimus: A Pharmacokinetic and Pharmacodynamic Phase I Study in Patients With Advanced Solid Tumours With an Expansion of Cohort With Patients With Recurrent/Metastatic Endometrial and Renal Cell Cancers
Brief Title: Gamma-Secretase/Notch Signalling Pathway Inhibitor RO4929097 and Temsirolimus in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02529; NCI-2011-02529 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 8500; CDR0000684714; PJC-005 (Other: University Health Network-Princess Margaret Hospital); 8500 (Other: CTEP); U01CA132123 (NIH)
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2013-10

CONDITIONS: Endometrial Papillary Serous Carcinoma; Recurrent Endometrial Carcinoma; Recurrent Renal Cell Cancer; Stage III Endometrial Carcinoma; Stage III Renal Cell Cancer; Stage IV Endometrial Carcinoma; Stage IV Renal Cell Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Endometrial Neoplasms; Carcinoma, Renal Cell | interventions — temsirolimus; Sirolimus; 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide

ARMS (1):
- Treatment (temsirolimus and RO4929097) (Experimental): Patients receive temsirolimus IV over 30 minutes on day -6 (course 1 only). Patients then receive temsirolimus IV or PO on days 1, 8, and 15 and gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: temsirolimus; Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: temsirolimus — Given IV or PO
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel
Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097 — Given PO
  Other Names: R4733; RO4929097
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of giving gamma-secretase/Notch signalling pathway inhibitor RO4929097 and temsirolimus together in treating patients with advanced solid tumors. Gamma-secretase/Notch signalling pathway inhibitor RO4929097 and temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose (RP2D) and safety profile of temsirolimus in combination with RO4929097 (gamma-secretase/Notch signalling pathway inhibitor RO4929097) in patients with advanced solid tumors.

SECONDARY OBJECTIVES:

I. To obtain pharmacokinetic (PK) profiles for both drugs when administered in combination in order to quantify the expected interactive effects in PK between these two agents.

II. To evaluate pharmacodynamic (PD) effects of both drugs when administered in combination, with the goal of identifying potential predictive and PD markers that need further exploration and validation in future trials.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive temsirolimus IV over 30 minutes on day -6 (course 1 only). Patients then receive temsirolimus IV or orally (PO) on days 1, 8, and 15 and gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Blood and tumor tissue samples may be collected periodically for pharmacokinetic and correlative analyses.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Meets one of the following sets of criteria:

  * Dose-escalation group:

    * Histologically and/or cytologically confirmed solid malignancy
    * Metastatic or unresectable disease
    * Disease for which standard curative or palliative measures do not exist or are no longer effective
  * Expansion group:

    * Histologically and/or cytologically confirmed endometrial (endometrioid, uterine papillary serious carcinoma, or carcinosarcoma) or renal cell cancer
    * Metastatic or unresectable disease
    * Disease for which standard curative or palliative measures do not exist or are no longer effective
* Measurable or non-measurable disease

  * Measurable disease is defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan
* No known brain metastases
* ECOG performance status (PS) 0-1 (Karnofsky PS 70-100%)
* Life expectancy > 12 weeks
* Leukocytes ≥ 3,000/mm^3
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 90 g/L (or ≥ 9 g/dL)
* Total bilirubin normal
* AST/ALT ≤ 2.5 times upper limit of normal
* Serum creatinine normal OR creatine clearance ≥ 60 mL/min
* Fasting cholesterol ≤ 350 mg/dL (9.0 mmol/L)
* Fasting triglycerides ≤ 400 mg/dL (4.56 mmol/L)
* No uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia or hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation

  * Note: it is acceptable to use corrected calcium when interpreting calcium levels
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use two effective forms of contraception (i.e., barrier contraception and one other method of contraception) for ≥ 4 weeks before, during, and for ≥ 12 months after completion of study therapy
* Able to swallow medication
* No malabsorption syndrome or other condition that would interfere with intestinal absorption
* No diarrhea ≥ grade 2 that is not under control with standard anti-diarrhea medications
* No uncontrolled concurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable anginal pectoris
  * Cardiac arrhythmia other than chronic, stable atrial fibrillation
  * Psychiatric illness or social situations that would limit compliance with study medications
* QTc ≤ 450 msec in males and a QTc ≤ 470 msec in females, as measured by ECG using Bazett formula
* No history of risk factors for QT interval prolongation including, but not limited to, a family or personal history of any of the following:

  * Long QT syndrome
  * Torsades de pointes
  * Recurrent syncope without known etiology
  * Sudden unexpected death
* No pre-existing significant pulmonary infiltrates of unknown origin
* No serologic positivity for hepatitis A, B, or C or history of liver disease or other forms of hepatitis or cirrhosis
* No HIV-positive patients on combination antiretroviral therapy
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to gamma-secretase inhibitor RO4929097 or temsirolimus
* Female patients may not donate ova during or after study treatment
* Male patients may not donate sperm during and for ≥ 12 months after completion of study treatment
* Patients may not donate blood during and for ≥ 12 months after completion of study treatment
* Any number of prior therapies allowed
* Recovered from side effects of previous systemic anticancer therapy to < CTCAE grade 2 toxicity (except alopecia)
* Concurrent leuteinizing hormone-releasing hormone agonist allowed in patients with castration-resistant prostate cancer
* No prior gamma-secretase inhibitor or any inhibitor of the PI3K/Akt/mTOR pathway
* At least 4 weeks since prior radiotherapy or systemic therapy (6 weeks for carmustine, nitrosoureas, or mitomycin C)

  * Exceptions may be made for low-dose, non-myelosuppressive radiotherapy for symptomatic palliation
* No other concurrent investigational agents
* No concurrent medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®)
* No concurrent medications that are strong inducers, inhibitors, or substrates of CYP3A4
* No antiarrhythmics or other concurrent medications with known potential to prolong QT interval
* No concurrent food that may interfere with the metabolism of gamma-secretase inhibitor RO4929097, including grapefruit or grapefruit juice
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-08; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose defined as the dose level at which less than or equal to 1 of 6 patients experienced DLT assessed using NCI CTCAE version 4.0 | 21 days
Safety profile assessed using NCI CTCAE version 4.0 | Up to 4 weeks post-treatment
  Frequency and severity of adverse events will be tabulated using counts and proportions detailing frequently occurring, serious and severe events of interest. Attempts to model associations between pharmacokinetic data with toxicity profiles will be performed primarily using descriptive statistics, however, logistic regression may be used if warranted.

SECONDARY OUTCOMES:
Objective response to treatment assessed using the RECIST criteria 1.1 | Up to 4 weeks post-treatment
  All analyses will be considered exploratory and inference will be performed with appropriate caution. For all statistical tests, two-sided tests will be performed and no p-value adjustment performed due to the exploratory nature of these tests. A p-value of 0.05 or less will be considered statistically significant.
Pharmacokinetic profiles | Pre-dose, 0.5, 1, 2, 4, 6 and 24 hours
  All analyses will be considered exploratory and inference will be performed with appropriate caution. For all statistical tests, two-sided tests will be performed and no p-value adjustment performed due to the exploratory nature of these tests. A p-value of 0.05 or less will be considered statistically significant.
Pharmacodynamic effects | Up to 4 weeks post-treatment
  All analyses will be considered exploratory and inference will be performed with appropriate caution. For all statistical tests, two-sided tests will be performed and no p-value adjustment performed due to the exploratory nature of these tests. A p-value of 0.05 or less will be considered statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (2):
- Canada (2):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario